CLINICAL TRIAL: NCT00528632
Title: Association of Gallbladder Cholesterolosis to Body Mass Index and Levels of Serum Cholesterol and Triglycerides.
Brief Title: Gallbladder Cholesterolosis, Body Mass Index and Serum Cholesterol and Triglycerides
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: MARCELO A. BELTRAN, MD, Hospital De La Serena
Other Study IDs: HLS-0012-09-07
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2009-07

CONDITIONS: Gallstones; Gallbladder Cholesterolosis
Keywords: Gallstones; Gallbladder; Cholesterolosis; Serum cholesterol; triglycerides; Body Mass Index
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cholesterolosis: I. Patients with gallbladder cholesterolosis and symptomatic cholelithiasis
  Interventions: Other: Specimen biopsy and serum laboratory tests
- Cholelithiasis: II. Patients without gallbladder cholesterolosis and with symptomatic cholelithiasis
  Interventions: Other: Specimen biopsy and serum laboratory tests

INTERVENTIONS:
Other: Specimen biopsy and serum laboratory tests — Biopsy of the surgical specimens (gallbladder) submitted after cholecystectomy
  Laboratory tests measuring levels of plasma total cholesterol and triglycerides

SUMMARY:
Cholesterolosis is a common finding in biopsy specimens of gallbladders surgically removed for cholelithiasis.

To the best of the investigators knowledge no study has analyzed the relationships of Body Mass Index, serum Cholesterol and Triglycerides and gallbladder cholesterolosis.

The purpose of this study is to analyze and find relations between gallbladder cholesterolosis, Body Mass Index, serum cholesterol and triglycerides.

DETAILED DESCRIPTION:
A prospective database including the following variables was filled out:

* Age
* Gender
* Diagnosis
* Weight
* Height
* Body Mass Index
* Histopathological results (Biopsy)
* Serum cholesterol
* Serum triglycerides

All elective patients older than 15 years of age submitted to cholecystectomy for symptomatic gallstones were included. Plasma cholesterol and triglycerides levels were measured 5 to 7 days before surgery. Only patients with chronic cholecystitis and with cholesterolosis according to the histology of the surgical specimen were included, we did not include any patient with acute cholecystitis or gallbladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients submitted to elective cholecystectomy
* Histopathological report of gallbladder cholesterolosis
* Histopathological report of chronic cholecystitis
* Patients older than 15 years of age

Exclusion Criteria:

* Patients younger than 15 years of age
* Pathological report missing from the hospital records

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients operated on elective basis for symtomatic gallbladder lithiasis
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A Beltran, MD, Principal Investigator — Hospital de La Serena; Carlos Barria, MD, Study Director — Hospital De La Serena - HISTOMED
Locations (1):
- Hospital De La Serena, La Serena, Coquimbo Region, Chile